CLINICAL TRIAL: NCT04846972
Title: Facilitate and Sustain Return to Work After Breast Cancer: Randomized Controlled Trial
Brief Title: Facilitate and Sustain Return to Work After Breast Cancer
Acronym: FASTRACS-RCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0536
Record Dates: First submitted 2021-04-14; First posted 2021-04-15 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer
Keywords: Work rehabilitation; Social psychology; Work psychology; Occupational health and medicine; Health program planning; Breast cancer; Work disability prevention; Intervention mapping
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: After inclusion, patients will receive standard care. Women allocated in this group will have the standard care.
- FASTRACS intervention group: Women allocated in the FASTRACS intervention group will follow a structured care pathway comprising three successive steps (end of chemotherapy interview with a nurse, transitional visit with their GP, pre-RTW visit with their OP), plus one optional step (late visit with an OP- RTW to work coordinator). Four tools will be used during the intervention (RTW guide or checklist for the patient, the GP, the OP and the employer).
  Interventions: Behavioral: FASTRACS intervention

INTERVENTIONS:
Behavioral: FASTRACS intervention — Intervention (4 steps) :
  * Penultimate to last chemotherapy : patient will receive tools of the intervention
  * 1 month after the end of oncological treatment (OT): patient will attend a general medicine consultation with the GP RTW checklist
  * 2 months after OT: patient will attend a pre RTW visit with the OP RTW checklist
  * 5 months after the end of OT: if the patient has not returned to work 10 months after inclusion, they will have a visit with an OP-RTW to work coordinator
  Self-questionnaires will evaluate quality of life (EORTC QLQC30, BR23, Euroqol (EQ-5D-5L)), anxiety and depression (HAD), employment status, self-efficacy to return to work (RTW-SE11), pre-RTW and RTW visit with the OP, social support, care consumption, physical activity (short IPAQ), perceived performance (WRF), work conditions. The implementation and use of the intervention tools will also be assessed: the patient guide, the employer guide, RTW checklists for the GP and the OP.
  Groups: FASTRACS intervention group

SUMMARY:
Breast cancer is the most frequent cancer in women in France, with an estimated 50,000 new cases each year. Prognosis is good, with a standardized survival rate of 85% at 5 years from diagnosis. Half of the women affected are of working age. Return to work after breast cancer faces barriers pertaining to the patients and their environment. There are social disparities in employment. Women with a lesser education and older women are at higher risk to lose their job. No intervention, to date, has demonstrated its effectiveness to facilitate return to work and reduce social disparities in employment after breast cancer. Current limitations of the interventions are to be over-medicalized and hospital-centered, to lack of theoretical foundations, and to be at risk of implementation failure. In a previous phase of the FASTRACS project, an intersectoral Community Advisory Board involving the different categories of stakeholders was launched to perform a needs analysis and build the logic model of the FASTRACS intervention with the Intervention Mapping protocol.

The main objective of the FASTRACS intervention is to facilitate sustained return to work (RTW) after breast cancer. Secondary objectives are to improve work-related quality of life and to decrease social disparities in employment after breast cancer.

Eligible patients are women: (1) aged between 18 and 55 years; (2) in paid employment; (3) diagnosed with a locally invasive non-metastatic first breast cancer (4) treated by surgery and chemotherapy in an adjuvant or neoadjuvant situation. Recruitment will take place in six investigating centres (centre hospitalier Lyon Sud, hôpital de la Croix-Rousse, hôpital femme-mère-enfant, centre Léon Bérard, hôpital Jean Mermoz, Clinique Charcot), after surgery and before the beginning of the chemotherapy. Women will be randomized between 2 groups (intervention vs control) with a stratification on the including centre, age, and socioprofessional category.

The intervention is founded on a multilevel logic model addressing the social determinants of health. It is composed of 4 successive steps during which 4 tools will be used. The first step involves an interview at the end of chemotherapy with a nurse, during which the patient is given a guide to returning to work. The second step is a transitional consultation in the month following the end of radiotherapy (or chemotherapy for patients without radiotherapy), with the general practitioner (GP), with a checklist designed to individualise the patient's care. The third step is a pre-RTW visit to the occupational physician (OP) at a time deemed appropriate by the patient and her GP, with a checklist to facilitate the accomodation of the workstation and the job retention strategy. The fourth and final step will only occur for patients who have not returned to work 10 months after inclusion, and will involve an interview with an OP specialised in return-to-work (RTW) coordination. The last tool is an employer's guide that will be given by the patient to her OP and her manager, with practical advice for managers and colleagues to facilitate the RTW process.

The evaluation of the intervention will be performed with mixed-methods by a realist randomized controlled trial including 210 patients in each group. For the effect evaluation, the primary outcome is a composite endpoint including: (a) a sustained return to work 12 months after oncological treatments (OT) ; and (b) the number of days on sick leave 12 months after oncological treatments. Secondary outcomes will include the patients' perspective (quality of life, anxiety, depression, RTW self-efficacy, social support, physical activity, work role functioning, work conditions), process outcomes (transition visit with the GP, pre RTW visit with the OP, other visits), and implementation outcomes (reach and use of the intervention tools).

Expected public health impact: Provided it is acceptable, effective and sustainable, the innovative intervention developed in this project is likely to decrease the impact of breast cancer on employment, and to decrease social disparities in employment after breast cancer. According to the mechanisms activated in each context under study (centres, workplaces), it could be scaled-up but also adapted to fit the needs of patients with other cancers or other chronic health conditions.

ELIGIBILITY:
Inclusion Criteria:

* Woman aged between 18 and 55
* With a diagnosis of invasive breast carcinoma of stage cTNM or pTNM I to III (UICC 8th edition), confirmed by histological examination
* Treated by intravenous cytotoxic chemotherapy in an adjuvant or neoadjuvant situation
* Breast surgery +/- of the axillary area, carried out within 3 months preceding the start of adjuvant chemotherapy, or scheduled after neo-adjuvant chemotherapy +/- radiotherapy.
* In salaried employment at the time of diagnosis (permanent or temporary contract, interim assignment, civil servant)
* Affiliated to a French social security scheme
* Reading, understanding and writing the French language
* Followed in one of the investigating centers
* Not opposing the collection of data

Exclusion Criteria:

* In situ carcinoma
* Distant metastases
* History or co-existence of another primary cancer (apart from a basal cell cancer of the skin and / or a non-mammary cancer in complete remission for more than 5 years)
* Recurrence or second breast cancer
* Without employment contract; self-employed or supported contract
* Cannot be followed for the duration of the study, for medical, social, family, geographic or psychological reasons
* Deprived of liberty by court or administrative decision

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women aged 18 to 55 with first invasive non-metastatic breast cancer (treated by surgery and chemotherapy in an adjuvant or neoadjuvant situation) and in paid employment at the time of diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2021-05-21 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
(a) a sustained return to work between inclusion and 12 months after oncological treatments; and (b) the number of days on sick leave between inclusion and 12 months after oncological treatments . | 12 months after oncological treatments (radiation therapy, or chemotherapy for patients without radiation therapy)
  The main analysis of the primary endpoint will be based on the net benefit of the intervention, estimated using the generalized pairwise comparison method

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - Hôpital Fleyriat, Bourg-en-Bresse
  - Hopital femme mère enfant, Hospices Civils de Lyon, Bron
  - Centre de lutte contre le Cancer JEAN PERRIN, CLERMONT-FERRAND, Clermont-Ferrand
  - Hopital de la croix rousse, Hospices Civils de Lyon, Lyon
  - Centre Léon Berard, Lyon
  - Hopital privé Jean Mermoz, Lyon
  - Service d'oncologie, Centre Hospitalier Annecy Genevois, Metz-Tessy
  - Hopital Lyon sud, Hospices civils de Lyon, Pierre-Bénite
  - Centre Hospitalo-universitaire de saint Etienne, Saint-Etienne
  - Clinique Charcot, Sainte-Foy-lès-Lyon
  - Centre Hospitalier de Valence, Valence

REFERENCES:
- [Derived] Fassier JB, Guittard L, Fervers B, Rouat S, Sarnin P, Carretier J, Broc G, Letrilliart L, Peron J, Lamort-Bouche M. Using intervention mapping to facilitate and sustain return-to work after breast cancer: protocol for the FASTRACS multicentre randomized controlled trial. BMC Cancer. 2024 Sep 5;24(1):1107. doi: 10.1186/s12885-024-12796-4. PMID 39237867